CLINICAL TRIAL: NCT02175446
Title: A Phase II Single Arm Trial Evaluating the Efficacy and Safety of Eribulin in Combination With Bevacizumab for 2-Line Treatment of HER 2-Negative Metastatic Breast Cancer Progressing After 1-Line Therapy With Bevacizumab and Paclitaxel
Brief Title: Safety and Efficacy Study of Eribulin in Combination With Bevacizumab for Second-line Treatment HER2- MBC Patients
Acronym: GIM11-BERGI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIM11-BERGI; 2013-003194-10 (EudraCT Number)
Record Dates: First submitted 2014-06-09; First posted 2014-06-26 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Metastatic Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
Keywords: Breast cancer; HER2Negative; Second line treatment; HER2-; MBC; Metastatic; Metastatic breast cancer; bevacizumab; eribulin; Human Epidermal Growth Factor Receptor 2-Negative
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental1 (Experimental): Bevacizumab and eribulin
  In this study all patients will receive:
  * Eribulin 1.23 mg/m2 on days 1, 8 every 3 weeks intravenously
  * Bevacizumab 15 mg/kg every 3 weeks intravenously or Bevacizumab 10 mg/kg every 2 weeks intravenously
  Interventions: Drug: Bevacizumab and eribulin

INTERVENTIONS:
Drug: Bevacizumab and eribulin — In this study, Bevacizumab and Eribulin are considered to be the "investigational study drugs". Bevacizumab is provided as 25 mg/ml concentrate for infusion. Vials contain 100 mg of Bevacizumab in 4 ml and/or 400 mg in 16 ml. Eribulin is provided as vials containing 1 mg/2 mL Eribulin as a 500 µg/mL solution in ethanol/water
  Other Names: Halaven; Avastin

SUMMARY:
In the second-line treatment setting for MBC, many agents, including antitubulin drugs (Taxanes, Vinorelbine) and antimetabolites (Capecitabine, Gemcitabine), have demonstrated activity, but no agent is clearly superior. Although some combinations of cytotoxic agents provide a small progression-free survival advantage, none has demonstrated an OS advantage, and toxicity is generally greater than for single agents. At present, there is no standard for this treatment setting. New treatments that could delay disease progression without systemic toxicity would represent a significant advancement.

DETAILED DESCRIPTION:
Metastatic breast cancer (MBC) is incurable, and the majority of patients succumb to their disease within 2 years of diagnosis.

Patients with MBC usually receive treatment with endocrine or cytotoxic chemotherapeutic agents, and treatment decisions are generally guided by the hormone receptor and Human Epidermal Growth Factor Receptor 2-Negative status of the disease, the number and location of metastases, and prior treatment history in both adjuvant and metastatic settings. In first- and second-line treatment settings of Metastatic Breast Cancer, numerous cytotoxic chemotherapy agents have demonstrated activity, including anti-tubulin drugs (Taxanes, Vinorelbine), Anthracyclines, and anti-metabolites (Capecitabine, Gemcitabine). However, no single agent has demonstrated a clear survival advantage over another, and use of sequential single-agent therapies is the most frequent approach. The choice of chemotherapy agent(s) is often determined by a number of factors, including history of prior therapy, treatment-free interval, and patient preference. Thus, no single standard treatment exists for patients with advanced disease. Patients who progress during or after their first treatment for Metastatic Brest Cancer typically have a short progression-free interval of 4-6 months and survive for 8-12 months. New treatment modalities are needed to improve clinical outcome and maintain the quality of life for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-specific procedures or treatment, as confirmation of the patient's awareness and willingness to comply with the study requirements.
* Female patients ≥18 years of age.
* Histologically confirmed Human Epidermal Growth Factor Receptor 2-Negative adenocarcinoma of the breast with documented progression of disease per investigator assessment following or during first-line treatment with Bevacizumab in combination with Paclitaxel for MBC; patients can have measurable or non-measurable disease. A minimum of 4 cycles of Bevacizumab 15 mg/kg or 6 cycles 10 mg/kg received in the first-line setting.
* Patients must have received Bevacizumab in combination with Paclitaxel as first line treatment. As part of their first line maintenance treatment, patients may have received:
* Bevacizumab monotherapy
* Bevacizumab in combination with endocrine treatment
* Nothing (for a period ≤ 6 weeks from the last Bevacizumab treatment)
* ECOG performance status (PS) of 0-2.
* At least 28 days since prior radiation therapy or surgery and recovery from treatment.
* Patients must have measurable disease which must be evaluable per RECIST v1.1.
* Estimated life expectancy of ≥12 weeks.

Exclusion Criteria:

Disease-specific exclusions

* Patients who have received anti-angiogenic therapy [e.g. tyrosine kinase inhibitors (TKIs) or anti-vascular endothelial growth factors (anti-VEGFs)] other than Bevacizumab for the first-line treatment of MBC.
* Patients who have exclusively received endocrine treatment in combination with Bevacizumab until the first progression.
* Positive or unknown Human Epidermal Growth Factor Receptor 2/neu status or for whom determination of Human Epidermal Growth Factor Receptor 2 status is not possible. In general, Human Epidermal Growth Factor Receptor 2 positive status will be identified by a FISH assay as evaluated at the institution, or, if FISH is unavailable, a 2+ or 3+ immunohistochemistry result (but method of identification may vary by region or institution).
* Current, recent (within 4 weeks or 2 half-lives, whichever is greater, before day 1) or planned participation in an experimental drug study - other than a Bevacizumab breast cancer study.
* Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix or breast within the last 5 years.
* Any laboratory values at baseline as described in the protocol;
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would prevent the patient from meeting the study requirements.
* Serious active infection requiring i.v. antibiotics and/or hospitalization at study entry.
* Patients who are treated with any medicinal product that contraindicates the use of any of the study drugs, may interfere with the planned treatment, affects patient compliance or puts the patient at high risk for treatment-related complications.

Bevacizumab-specific exclusions: (see protocol)

Eribulin-specific exclusions: (see protocol)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 30 months
  ORR will be evaluated for those patients who have a response to second-line treatment as defined per RECIST version 1.1 in patients with measurable disease according to RECIST version 1.1. ORR will be based on the best overall response (BOR) as defined by RECIST Guidelines v. 1.1.

SECONDARY OUTCOMES:
Progression free survival | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 30 months
  Second-line progression-free survival, defined as the time from first dosing to the first documented disease progression or death from any cause, whichever occurs first.
Overall Survival | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 30 months
  OS is defined as the time from first dosing in second line to death from any cause.
Clinical Benefit Rate | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 30 months
  Clinical Benefit Rate is the proportion of patients with a complete or partial response or with stable disease at 24 weeks.
Duration of response | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 30 months
  Duration of response measures the length of the response in those patients who responded to treatment.
Safety | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 30 months
  Safety of second line treatment will be evaluated by the frequency of AEs and SAEs, cardiac events, clinically significant abnormal laboratory tests, vital signs, and ECOG PS. All patients who received at least one dose of study treatment will be included in the safety analysis.
Quality of life | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 30 months
  QoL and symptom control will be assessed using the FACT-B questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Grazia Arpino, MD, Principal Investigator — Dipartimento di Medicina Clinica e Chirurgia Oncologia Università degli Studi di Napoli "Federico II"
Locations (17):
- Italy (17):
  - Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona
  - Ospedale 'F. Spaziani', Frosinone
  - I.R.C.C.S. A.O.U. San Martino - I.S.T., Genova
  - Ospedale Unico Versilia, Lido di Camaiore
  - Ospedale San Luca Istituto Tumori Toscano, Lucca
  - Ospedale civile di Macerata, Macerata
  - A.O.R.N. "A. Cardarelli", Naples
  - Università degli Studi di Napoli "Federico II", Naples
  - Istituto Nazionale Tumori - IRCCS "Fondazione G.Pascale", Napoli
  - AORN - Ospedali dei Colli Monaldi-Cotugno - C.T.O., Napoli
  - I.R.C.C.S. Fondazione Salvatore Maugeri, Pavia
  - Azienda Ospedaliera Universitaria Pisana - Ospedale S. Chiara, Pisa
  - Presidio Ospedaliero Felice Lotti Pontedera, Pontedera
  - Istituto Regina Elena per lo studio e la cura dei tumori, Roma
  - Azienda Ospedaleira Universitaria San Giovanni di Dio e Ruggi d'aragona, Salerno
  - Ospedale 'SS. Trinità', Sora
  - Azienda Ospedaliera Universitaria Santa Maria della Misericordia di Udine, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen A, et al. Clinical outcomes in Bevacizumab (BV)-treated patients (pts) with metastatic colorectal cancer (mCRC): Results from ARIES observational cohort study (OCS) and confirmation of BRITE data on BV beyond progression (BBP). ASCO 2010
- [Background] Saab TB, et al. Bevacizumab (BV) plus chemotherapy (CT) in 2nd line metastatic colorectal cancer (mCRC): Initial results from ARIES a second observational cohort study. ASCO 2010.
- [Result] Greenberg PA, Hortobagyi GN, Smith TL, Ziegler LD, Frye DK, Buzdar AU. Long-term follow-up of patients with complete remission following combination chemotherapy for metastatic breast cancer. J Clin Oncol. 1996 Aug;14(8):2197-205. doi: 10.1200/JCO.1996.14.8.2197. PMID 8708708
- [Result] Chia SK, Speers CH, D'yachkova Y, Kang A, Malfair-Taylor S, Barnett J, Coldman A, Gelmon KA, O'reilly SE, Olivotto IA. The impact of new chemotherapeutic and hormone agents on survival in a population-based cohort of women with metastatic breast cancer. Cancer. 2007 Sep 1;110(5):973-9. doi: 10.1002/cncr.22867. PMID 17647245
- [Result] Hamilton A, Hortobagyi G. Chemotherapy: what progress in the last 5 years? J Clin Oncol. 2005 Mar 10;23(8):1760-75. doi: 10.1200/JCO.2005.10.034. No abstract available. PMID 15755984
- [Result] Perez EA. Impact, mechanisms, and novel chemotherapy strategies for overcoming resistance to anthracyclines and taxanes in metastatic breast cancer. Breast Cancer Res Treat. 2009 Mar;114(2):195-201. doi: 10.1007/s10549-008-0005-6. Epub 2008 Apr 29. PMID 18443902
- [Result] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Result] Inai T, Mancuso M, Hashizume H, Baffert F, Haskell A, Baluk P, Hu-Lowe DD, Shalinsky DR, Thurston G, Yancopoulos GD, McDonald DM. Inhibition of vascular endothelial growth factor (VEGF) signaling in cancer causes loss of endothelial fenestrations, regression of tumor vessels, and appearance of basement membrane ghosts. Am J Pathol. 2004 Jul;165(1):35-52. doi: 10.1016/S0002-9440(10)63273-7. PMID 15215160
- [Result] Baffert F, Le T, Sennino B, Thurston G, Kuo CJ, Hu-Lowe D, McDonald DM. Cellular changes in normal blood capillaries undergoing regression after inhibition of VEGF signaling. Am J Physiol Heart Circ Physiol. 2006 Feb;290(2):H547-59. doi: 10.1152/ajpheart.00616.2005. Epub 2005 Sep 19. PMID 16172161
- [Result] Kamba T, Tam BY, Hashizume H, Haskell A, Sennino B, Mancuso MR, Norberg SM, O'Brien SM, Davis RB, Gowen LC, Anderson KD, Thurston G, Joho S, Springer ML, Kuo CJ, McDonald DM. VEGF-dependent plasticity of fenestrated capillaries in the normal adult microvasculature. Am J Physiol Heart Circ Physiol. 2006 Feb;290(2):H560-76. doi: 10.1152/ajpheart.00133.2005. Epub 2005 Sep 19. PMID 16172168
- [Result] Mancuso MR, Davis R, Norberg SM, O'Brien S, Sennino B, Nakahara T, Yao VJ, Inai T, Brooks P, Freimark B, Shalinsky DR, Hu-Lowe DD, McDonald DM. Rapid vascular regrowth in tumors after reversal of VEGF inhibition. J Clin Invest. 2006 Oct;116(10):2610-21. doi: 10.1172/JCI24612. PMID 17016557
- [Result] Miller KD, Chap LI, Holmes FA, Cobleigh MA, Marcom PK, Fehrenbacher L, Dickler M, Overmoyer BA, Reimann JD, Sing AP, Langmuir V, Rugo HS. Randomized phase III trial of capecitabine compared with bevacizumab plus capecitabine in patients with previously treated metastatic breast cancer. J Clin Oncol. 2005 Feb 1;23(4):792-9. doi: 10.1200/JCO.2005.05.098. PMID 15681523
- [Result] Gray R, Bhattacharya S, Bowden C, Miller K, Comis RL. Independent review of E2100: a phase III trial of bevacizumab plus paclitaxel versus paclitaxel in women with metastatic breast cancer. J Clin Oncol. 2009 Oct 20;27(30):4966-72. doi: 10.1200/JCO.2008.21.6630. Epub 2009 Aug 31. PMID 19720913
- [Result] Miles DW, Chan A, Dirix LY, Cortes J, Pivot X, Tomczak P, Delozier T, Sohn JH, Provencher L, Puglisi F, Harbeck N, Steger GG, Schneeweiss A, Wardley AM, Chlistalla A, Romieu G. Phase III study of bevacizumab plus docetaxel compared with placebo plus docetaxel for the first-line treatment of human epidermal growth factor receptor 2-negative metastatic breast cancer. J Clin Oncol. 2010 Jul 10;28(20):3239-47. doi: 10.1200/JCO.2008.21.6457. Epub 2010 May 24. PMID 20498403
- [Result] Robert NJ, Dieras V, Glaspy J, Brufsky AM, Bondarenko I, Lipatov ON, Perez EA, Yardley DA, Chan SY, Zhou X, Phan SC, O'Shaughnessy J. RIBBON-1: randomized, double-blind, placebo-controlled, phase III trial of chemotherapy with or without bevacizumab for first-line treatment of human epidermal growth factor receptor 2-negative, locally recurrent or metastatic breast cancer. J Clin Oncol. 2011 Apr 1;29(10):1252-60. doi: 10.1200/JCO.2010.28.0982. Epub 2011 Mar 7. PMID 21383283
- [Result] Brufsky AM, Hurvitz S, Perez E, Swamy R, Valero V, O'Neill V, Rugo HS. RIBBON-2: a randomized, double-blind, placebo-controlled, phase III trial evaluating the efficacy and safety of bevacizumab in combination with chemotherapy for second-line treatment of human epidermal growth factor receptor 2-negative metastatic breast cancer. J Clin Oncol. 2011 Nov 10;29(32):4286-93. doi: 10.1200/JCO.2010.34.1255. Epub 2011 Oct 11. PMID 21990397
- [Result] Grothey A, Sugrue MM, Purdie DM, Dong W, Sargent D, Hedrick E, Kozloff M. Bevacizumab beyond first progression is associated with prolonged overall survival in metastatic colorectal cancer: results from a large observational cohort study (BRiTE). J Clin Oncol. 2008 Nov 20;26(33):5326-34. doi: 10.1200/JCO.2008.16.3212. Epub 2008 Oct 14. PMID 18854571
- [Result] Bennouna J, Sastre J, Arnold D, Osterlund P, Greil R, Van Cutsem E, von Moos R, Vieitez JM, Bouche O, Borg C, Steffens CC, Alonso-Orduna V, Schlichting C, Reyes-Rivera I, Bendahmane B, Andre T, Kubicka S; ML18147 Study Investigators. Continuation of bevacizumab after first progression in metastatic colorectal cancer (ML18147): a randomised phase 3 trial. Lancet Oncol. 2013 Jan;14(1):29-37. doi: 10.1016/S1470-2045(12)70477-1. Epub 2012 Nov 16. PMID 23168366
- [Result] Cigler T, Vahdat LT. Eribulin mesylate for the treatment of breast cancer. Expert Opin Pharmacother. 2010 Jun;11(9):1587-93. doi: 10.1517/14656566.2010.486790. PMID 20450446
- [Result] Kuznetsov G, Towle MJ, Cheng H, Kawamura T, TenDyke K, Liu D, Kishi Y, Yu MJ, Littlefield BA. Induction of morphological and biochemical apoptosis following prolonged mitotic blockage by halichondrin B macrocyclic ketone analog E7389. Cancer Res. 2004 Aug 15;64(16):5760-6. doi: 10.1158/0008-5472.CAN-04-1169. PMID 15313917
- [Result] Vahdat LT, Pruitt B, Fabian CJ, Rivera RR, Smith DA, Tan-Chiu E, Wright J, Tan AR, Dacosta NA, Chuang E, Smith J, O'Shaughnessy J, Shuster DE, Meneses NL, Chandrawansa K, Fang F, Cole PE, Ashworth S, Blum JL. Phase II study of eribulin mesylate, a halichondrin B analog, in patients with metastatic breast cancer previously treated with an anthracycline and a taxane. J Clin Oncol. 2009 Jun 20;27(18):2954-61. doi: 10.1200/JCO.2008.17.7618. Epub 2009 Apr 6. PMID 19349550
- [Result] Cortes J, Vahdat L, Blum JL, Twelves C, Campone M, Roche H, Bachelot T, Awada A, Paridaens R, Goncalves A, Shuster DE, Wanders J, Fang F, Gurnani R, Richmond E, Cole PE, Ashworth S, Allison MA. Phase II study of the halichondrin B analog eribulin mesylate in patients with locally advanced or metastatic breast cancer previously treated with an anthracycline, a taxane, and capecitabine. J Clin Oncol. 2010 Sep 1;28(25):3922-8. doi: 10.1200/JCO.2009.25.8467. Epub 2010 Aug 2. PMID 20679609
- [Result] Twelves C, Cortes J, Vahdat LT, Wanders J, Akerele C, Kaufman PA. Phase III trials of eribulin mesylate (E7389) in extensively pretreated patients with locally recurrent or metastatic breast cancer. Clin Breast Cancer. 2010 Apr;10(2):160-3. doi: 10.3816/CBC.2010.n.023. PMID 20299316
- [Result] Cortes J, O'Shaughnessy J, Loesch D, Blum JL, Vahdat LT, Petrakova K, Chollet P, Manikas A, Dieras V, Delozier T, Vladimirov V, Cardoso F, Koh H, Bougnoux P, Dutcus CE, Seegobin S, Mir D, Meneses N, Wanders J, Twelves C; EMBRACE (Eisai Metastatic Breast Cancer Study Assessing Physician's Choice Versus E7389) investigators. Eribulin monotherapy versus treatment of physician's choice in patients with metastatic breast cancer (EMBRACE): a phase 3 open-label randomised study. Lancet. 2011 Mar 12;377(9769):914-23. doi: 10.1016/S0140-6736(11)60070-6. Epub 2011 Mar 2. PMID 21376385
- [Result] von Minckwitz G, du Bois A, Schmidt M, Maass N, Cufer T, de Jongh FE, Maartense E, Zielinski C, Kaufmann M, Bauer W, Baumann KH, Clemens MR, Duerr R, Uleer C, Andersson M, Stein RC, Nekljudova V, Loibl S. Trastuzumab beyond progression in human epidermal growth factor receptor 2-positive advanced breast cancer: a german breast group 26/breast international group 03-05 study. J Clin Oncol. 2009 Apr 20;27(12):1999-2006. doi: 10.1200/JCO.2008.19.6618. Epub 2009 Mar 16. PMID 19289619
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774